CLINICAL TRIAL: NCT06783816
Title: A Multicenter, Single Arm, Open Label Clinical Study on the Novel CAR-T Combined Expression of IL-15 in the Treatment of Malignant Hematological Tumors
Brief Title: A Novel CAR-T Combined Expression of IL-15 in the Treatment of Malignant Hematological Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VC-HM-001
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-03

CONDITIONS: Acute Lymphocytic Leukemia; Lymphoma,Non-Hodgkin; Relapsed Refractory Multiple Myeloma
Keywords: CAR-T; IL-15; malignant hematological tumors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group1 (Experimental): In patients with acute B-lymphoblastic leukemia, the dose was 0.5-1.5×10^6 CAR-positive T cells /kg body weight. The usual dose of B-cell non-Hodgkin lymphoma was 0.5-2.0 ×10^6/kg CAR-positive T cells. The initial dose of r/r multiple myeloma is 1x10^6/kg, and the dose of 3x10^6/kg and 5x10^6/kg are generally proposed to increase successively.
  Interventions: Drug: chimeric antigen receptor gene modified T cells

INTERVENTIONS:
Drug: chimeric antigen receptor gene modified T cells — The rate of intravenous infusion of CAR T cells was 10 mL to 20 mL/min, and the infusion was performed using a blood transfusion apparatus with a filter screen. Use saline rinsing tube prior to infusion; Rinse the infusion bag with 10 mL~30 mL normal saline.

SUMMARY:
The is a multicenter, single arm, open label clinical study on the novel CAR-T combined expression of IL-15 in the treatment of malignant hematological tumors.Plan to recruit 45 subjects with malignant hematological tumors.

DETAILED DESCRIPTION:
The main objective is to evaluate the safety and efficacy of a novel CAR-T therapy that co expresses IL-15 in malignant hematological tumors.

The secondary objective is to investigate the in vivo survival time of the novel CAR-T co expressing IL-15 and the activation and proliferation of a novel CAR-T co expressing IL-15 in vivo.

ELIGIBILITY:
Inclusion Criteria:

* I (or the authorized representative/legal guardian) agree and have signed an informed consent form, and am willing and capable of following the planned visits, research treatments, laboratory tests, and other research procedures;
* Histopathological or flow cytometric diagnosis of CD19 and/or CD22, BCMA-positive hematological malignancies;

  -≥15 years old, ≤80 years old;
* If you meet one of the following three conditions, you can be included in the group:-Patients with recurrent or refractory hematologic malignancies treated with one standard chemotherapy regimen and one salvage regimen;-Minimal residual lesions persist after treatment with one standard chemotherapy regimen and one salvage regimen;-Patients with recurrence after hematopoietic stem cell transplantation;
* Estimated survival ≥12 weeks;
* Good heart, liver and kidney function:
* Serum creatinine ≤ 1.5 mg/dL (1mg/dl=88.4umol/L); Serum ALT/AST ≤ 2.5 ULN; Total bilirubin ≤ 1.5 mg/dl (1mg/dl=17.1umol/L):
* Cardiac ejection fraction ≥50%, cardiac ultrasound showed centropericardial effusion:
* Eastern Oncology Collaborative Group Activity Status Score (ECOG)0-3;
* Able to understand and voluntarily sign informed consent; If the subject is a child, the guardian will sign the informed consent.

If the answer to any of the above is "no", the subject will not be allowed to participate in this study.

Exclusion Criteria:

* Have a New York Heart Association (NYHA) classification > Class III heart failure or myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically prominent heart disease within one year prior to signing the consent form, or have a QTC interval >480ms at the time of screening (QTC interval is calculated using the Fridericia formula);
* Have active GVHD, or need immunosuppressants;
* Other malignancies were present within 5 years prior to screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, and breast ductal carcinoma in situ after radical resection of local prostate cancer;
* The presence of an active or uncontrolled infection requiring systemic treatment (except for mild genitourinary and upper respiratory tract infections) in the 7 days prior to screening;
* If HBSAg or HbCAb positive peripheral blood hepatitis B virus (HBV)DNA is higher than the lower limit of detection, it should be excluded. If hepatitis C virus (HCV) antibody positive, peripheral blood HCVRNA positive should be excluded; (HIV) antibody-positive; -Cytomegalovirus (CMV)DNA test positive for human immunodeficiency virus; Those who test positive for Treponema pallidum specific antibody (TPPA) should be excluded;
* Participating in another clinical trial within 4 weeks prior to the signing of the informed consent, or the signing date of the informed consent is still within 5 half-lives of the drug (whichever is longer) since the last drug used in the last clinical trial;
* A history of severe allergy to biological products;
* Systemic diseases that are considered unstable by the investigator: including but not -limited to severe liver, kidney, or metabolic diseases requiring medical treatment;
* Pregnant or lactating women, and female subjects who plan pregnancy within 2 years after cell transfusion or male subjects whose partner plans pregnancy within 2 years after cell transfusion;
* Conditions that the investigator believes may increase the risk to the subject or interfere with the test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
monitor the survival time of CAR-T in vivo | 6 months
  The survival of CAR-T in vivo will be monitored periodically by flow cytometry after CAR T reinfusion.
Record antitumor effects after reinfusion of CAR-T | 28 days
  Determine partial response (PR) or complete response (CR) for subjects with active disease. In view of the small number of subjects, remission should be recorded in detail; For subjects treated with minimal residual lesion (MRD), MRD clearance results were recorded.

SECONDARY OUTCOMES:
Disease-free survival | 3 years
  DFS was calculated from the first CAR-T cell infusion to death, progression of the disease, relapse or gene recurrence, whichever came first, or last visit.
Overall Survival | 3 years
  OS was calculated from the first CAR-T cell infusion to death or last follow-up

OTHER OUTCOMES:
The copy number of CAR-T cells | 12 months
  The copy number of CAR-T cells amplified in peripheral blood after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China